CLINICAL TRIAL: NCT01250808
Title: Technology Platform and System Construction of Clinical Evaluation Studies on New Drugs of Hematological Malignancy
Status: Available | Type: Expanded Access
Sponsor: Peking University (Other)
Responsible Party: Huang Xiaojun, Institute of Hematology, Peking University.
Other Study IDs: 2008ZX09312-026
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

INTERVENTIONS:
Drug: Bortezomib/Dexamethasone/Melphalan — Induction therapy: The treatment will continue for 3-4 cycles and each cycle will be last 21 days.
  Bortezomib 1.3mg/m2, twice weekly for two weeks (days 1, 4, 8, and 11) of each cycle + Dexamethasone 20mg/m2, on days 1-4 of each cycle.
  Bortezomib 1.0mg/m2, twice weekly for two weeks (days 1, 4, 8, and 11) of each cycle + Dexamethasone 20mg/m2, on days 1-4 of each cycle.
  Bortezomib 1.6mg/m2, once weekly for two weeks (days 1, 8) of each cycle + Dexamethasone 20mg/m2, on days 1-4 of each cycle and on days 9-12 of the first and second cycles.
  ASCT therapy:
  Melphalan 200mg/m2 +Bortezomib 1.0mg/m2 for four times. Melphalan 200mg/m2 +Bortezomib 1.0mg/m2 for two times.

SUMMARY:
Multiple Myeloma (MM) is the second diagnosed malignancy of hematological malignancies. The previous study pointed out that the dosage and course of Bortezomib including the dose of concomitant drugs used to treatment MM patients did not get the preferred treatment program, so we are going to determine the optimal doses and course of Bortezomib through the prospective, multicenter clinical trial and evaluate the efficiency and safety of different program.

ELIGIBILITY:
Inclusion Criteria:

1. Obtain informed consent form (ICF) signed by patients or its relative.
2. Patients newly diagnosed multiple myeloma (MM). (Not include patients with multiple solitary extramedullary plasmacytoma and those atⅠstage of Durie-Salmon staging system)
3. Measurable serum protein:

   IgG type of MM: serum M-protein≥ 1.0g/dl or urine M-protein≥ 200mg/24h. IgA type of MM: serum M-protein≥0.5g/dl or urine M-protein≥200mg/24h. IgM type of MM: (IgM M-protein and osteolytic lesion showed in X-ray):serum protein≥ 1.0g/dl or urine M-protein≥ 200mg/24h. IgD type of MM: serum M-protein≥0.05g/dl or urine M-protein≥200mg/24h. Light chain type of MM: serum M-protein≥ 1.0g/dl or urine M-protein≥ 200mg/24h.
4. Physical score 0~2 grade(WHO standard), and able to comply with the visit time and protocol requirements.

Exclusion Criteria:

1. Diagnosed with relapsed multiple myeloma.
2. Any serious diseases which may lead patients suffer from unaccepted risk.
3. Female patients who is pregnant or breast-feeding.
4. Histories of other malignant tumors other than MM, except those patients whose disease have been cured for at least 3 years. Exception: basal-cell carcinoma, squamous cell carcinoma, carcinoma in situ of uterine cervix, breast carcinoma in situ,occasionally prostatic cancer histological discovery(at stage T1a or T1B defined as TNM classification).
5. Not be able to understand or comply with the investigate protocol.
6. Patients with grade 2 or higher peripheral neuropathy before treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology,Peking University, Beijing, China